CLINICAL TRIAL: NCT05787340
Title: Investigation From Biopsychosocial Perspective of Patients With Rheumatic Disease With Covid-19 Who Participated in a Biopsychosocial Exercise Program: A Case Series With 6-Month Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Nazli Elif Nacar, Physiotherapist (MSc), Kahramanmaras Sutcu Imam University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kahramanmaras S I U
Record Dates: First submitted 2022-11-26; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Rheumatic Diseases
Keywords: Cognitive Exercise Therapy Approach; biopsychosocial exercise; rheumatology rehabilitation; qualitative research; case report
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BETY exercise group (Experimental): intervention group Bilişsel Egzersiz Terapi Yaklaşımı (BETY, Cognitive Exercise Therapy Approach) is a group exercise method that conforms to the biopsychosocial model via telerehabilitation
  Exercise dosage is 60 minute three days a week.
  Interventions: Other: Bilişsel Egzersiz Terapi Yaklaşımı (BETY, Cognitive Exercise Therapy Approach)

INTERVENTIONS:
Other: Bilişsel Egzersiz Terapi Yaklaşımı (BETY, Cognitive Exercise Therapy Approach) — Bilişsel Egzersiz Terapi Yaklaşımı (BETY, Cognitive Exercise Therapy Approach) is a group exercise method that conforms to the biopsychosocial model via telerehabilitation.

SUMMARY:
Objective: This novel study aimed to interrogate from a biopsychosocial perspective the health conditions during the Covid-19 infection and long-Covid periods of 5 patients with rheumatic disease infected with Covid-19 who had acquired the habit of regular exercise before the pandemic.

Method: This case study included five patients suffering from Covid-19 infection among patients with rheumatic disease who had acquired the habit of regular exercise before the Covid-19 pandemic. It was applied a questionnaire to the patients from a biopsychosocial perspective to see the short and long-term effects of Covid-19 during and after quarantine. Moreover, the study used the BETY-Biopsychosocical Questionnaire (BETY-BQ) to evaluate a biopsychosocial point, Health Assessment Questionnaire (HAQ) to measure functional status, and the Hospital Anxiety and Depression Scale (HADS) to assess anxiety and depression.

Results: In BETY-BQ, HAQ, and HADS, there was an unfavorable increase in overall scores of all patients during Covid-19. After six months, although the results from these three scales improved, some of the patients could not return to their pre-covid state.

Conclusions: The patients participating in the telerehabilitation were able to return to everyday life after Covid more efficiently and overcome post-Covid symptoms easily. This study is important in guiding the exercise approach for patients with rheumatic diseases in pandemics such as Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the rheumatic disease passed for at least six months after their Covid-19 infection between the ages of 18-65 were included in the study.

Exclusion Criteria:

* Exclusion criteria were the presence of deformity that does not allow exercise, cardiopulmonary disorders, uncontrolled endocrine system diseases, severe psychiatric illnesses, and insufficient skills in using a smartphone.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Qualitative research | at 6 month
  We aimed to complete qualitative interviews to investigate the biopsychosocial perspectives of patients with rheumatic diseases in the study. A team of four physiotherapists experienced in rheumatic diseases prepared an interview guide based on prior studies in the literature. The interview guide consisted of 25-item questions from a biopsychosocial perspective to see the short and long-term effects of Covid-19 infection on these patients during and after quarantine.

SECONDARY OUTCOMES:
Bilişsel Egzersiz Terapi Yaklaşımı-Biopsychosocial Questionnaire (BETY-BQ) | before infection, during infection and at 6 month after infection
  The scale consists of 30 items. The scoring of the scale was made using a 5-point Likert system. Each question is scored as "No never: 0 Yes rarely: 1 Yes sometimes: 2 Yes often: 3 Yes always: 4" and gives a total score over 30 items. A high score means that the biopsychosocial situation is 'bad'.
Health Assessment Questionnaire (HAQ) | before infection, during infection and at 6 month after infection
  The functional status of the patients was determined by the Health Assessment Questionnaire. The 20-question scale has 8 subtitles that include dressing, sitting, eating, walking, hygiene, reaching out, grasping, and daily life activities. Each answer is scored between 0 and 3 points. It means "0 = Without difficulty, 1 = A little difficult, 2 = Very difficult and 3 = I can never do it". The total score is the average score derived from 8 points for each category.High score indicates low functional status.
Hospital Anxiety and Depression Scale (HADS) | before infection, during infection and at 6 month after infection
  The anxiety and depression of the patients was determined by Hospital Anxiety and Depression Scale (HADS). This questionnaire is consisting of 14 questions with 4 options. The higher the score, the higher the anxiety and depression levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Nazli Elif Nacar, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No